CLINICAL TRIAL: NCT00847444
Title: Simultaneous Study of Docetaxel Based Anthracycline Free Adjuvant Treatment Evaluation, as Well as Life Style Intervention Strategies
Brief Title: Docetaxel Based Anthracycline Free Adjuvant Treatment Evaluation, as Well as Life Style Intervention
Acronym: SUCCESS-C
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Philip Hepp (Other)
Responsible Party: Sponsor-Investigator, Philip Hepp, Sponsors Representant, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUCCESS-C Trial
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AA (Active Comparator): Drug intervention
  Interventions: Drug: Drug-based intervention
- BA (Active Comparator): Lifestyle intervention
  Interventions: Behavioral: Lifestyle-based Intervention
- BB (No Intervention): No individualized lifestyle intervention program.

INTERVENTIONS:
Drug: Drug-based intervention — Randomization A AA: 3 cycles of 5-Fluorouracil 500 mg/m² i.v. body surface area and Epirubicine 100 mg/m² i.v. and Cyclophosphamide 500 mg/m² i.v., (FEC100), each administered on day 1, repeated on day 22, subsequently followed by 3 cycles of Docetaxel 100 mg/m² body surface area i.v. (D), administered on day 1, repeated on day 22 AB: 6 cycles of Docetaxel 75 mg/m² and Cyclophosphamide 600 mg/m² i.v. body surface area i.v. (DC), administered on day 1, repeated on day 22
  Arms: AA
Behavioral: Lifestyle-based Intervention — All Patients with a Body Mass Index (BMI) of 24 - 40 kg/m² at the time of enrollment will be subsequently randomized as follows:
  Second randomization B BA: Lifestyle intervention program to reduce body weight comprising individual weight loss, diet and physical activity goals in the framework of a 2-year standardized and structured telephone and mail-based intervention.
  Arms: BA

SUMMARY:
This is an open-label, multicenter, 2x2 factorial design, randomized controlled, Phase III study comparing the disease free survival after randomisation in patients treated with 3 cycles of Epirubicine-Fluorouracil-Cyclophosphamide(FEC)-chemotherapy, followed by 3 cycles of Docetaxel(D)-chemotherapy, versus 6 cycles of Docetaxel- Cyclophosphamide (DC)-chemotherapy, and to compare the disease free survival in patients with BMI of 24 - 40 kg/m² after randomisation with versus without the lifestyle intervention. Patients will be required to have histopathological proof of a HER2/neu negative tumor and: axillary lymph node metastases (pN1-3) or high risk node negative, defined as: 'pT ≥2 or histopathological grade 3, or age ≤35 or negative hormone receptor status, but are not allowed to have evidence of distant disease. Patients will have to be entered into the study no later than 6 weeks after complete resection of the primary tumor. No other antineoplastic treatment other than surgical treatment, the defined cytotoxic and endocrine treatment and radiotherapy will be allowed prior to study entry and during the course of the study.

DETAILED DESCRIPTION:
Rationale:

* Taxane based chemotherapy will be established as treatment standard in the adjuvant setting of early breast cancer
* 3xFEC100, followed by 3xDoc100 has been established as standard treatment option for node-positive breast cancer
* Anthracycline based regimens do not seem to be superior in Her2/neu-negative patients (Gennari et al., Slamon et al.)
* Dietary intervention can improve outcome in patients with early breast cancer (WINS, Chlebowski et al.)

Primary Endpoints:

* The first primary objective of this study is to compare disease free survival after randomisation in patients treated with a combination of 5-FU/Epirubicine/Cyclophosphamide followed by Docetaxel vs. Docetaxel/Cyclophosphamide
* The second primary objective of this study is to compare disease free survival after randomisation in patients with vs. without lifestyle intervention

Design:

Prospectively randomized open label Phase III study with 2x2 factorial design

ELIGIBILITY:
Patients may be included in the study only if they meet all the following criteria:

1. Primary epithelial invasive carcinoma of the breast pT1-4, pN0-3, pM0
2. No evidence of HER2/neu overexpressing (IHC neg or +) or amplifying (FISH neg.) tumor
3. Histopathological proof of axillary lymph node metastases (pN1-3) or high risk node negative, defined as at least one criterion of the following: 'pT ≥2, histopathological grade 3, age ≤35, negative hormone receptor'
4. Complete resection of the primary tumor with margins of resection free of invasive carcinoma not more than 6 weeks ago
5. Females ≥ 18 years of age
6. Performance status ≤ 2 on ECOG-Scale
7. Adequate bone marrow reserve: leucocytes ≥ 3.0 x 109/l and platelets ≥ 100 x 109/l
8. Bilirubin within the reference laboratory's normal range, ASAT (SGOT), ALAT (SGPT) and AP within 1,5 fold of the reference laboratory's normal range for patients
9. Willingness to participate in a telephone-based lifestyle intervention programme [10.] Intention of regular follow up visits for the duration of the study [11.] Ability to understand the nature of the study and to give written informed consent

Patients will be excluded from the study for any of the following reasons:

1. Inflammatory breast cancer
2. Previous or concomitant cytotoxic or other systemic antineoplastic treatment which is not part of this study
3. A second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin)
4. Cardiomyopathy with impaired ventricular function (NYHA > II), cardiac arrhythmias influencing LVEF and requiring medication, history of myocardial infarction or angina pectoris within the last 6 months, or arterial hypertension not being controlled by medication
5. Any known hypersensitivity against Docetaxel, Epirubicine, Cyclophosphamide, or any other medication included in the study protocol. The contraindication, warning notices and measures of precaution of the products, as notified in the product infroamtion, have to be respected
6. Use of any investigational agent within 3 weeks prior to inclusion
7. Patients in pregnancy or breast feeding (in premenopausal women anticonception has to be assured)
8. Insulin-requiring diabetes mellitus (non-insulin requiring patients with type 2 diabetes are eligible for the study)
9. Serious digestive and/or absorptive problems that exclude adherence to the study diet [10.] Self-reported inability to walk at least one kilometer (at any pace) [11.] Cardiovascular, respiratory or musculoskeletal disease or joint problems that preclude moderate physical activity. Moderate arthritis that does not preclude physical activity is not a reason for exclusion [12.] Psychiatric disorders or conditions that would preclude participation in the study intervention [13.] Patients not sufficiently fluent in German language to understand the nature of this study and any of the interventional measures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3547 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-09 (Actual); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
The first primary objective of this study is to compare disease free survival after randomisation in patients treated with a combination of 5-FU/Epirubicine/Cyclophosphamide followed by Docetaxel vs. Docetaxel/Cyclophosphamide | 60 months

SECONDARY OUTCOMES:
The second primary objective of this study is to compare disease free survival after randomisation in patients with vs. without lifestyle intervention | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Janni, Prof. Dr. med., Study Director — Klinikum der Heinrich-Heine-Universität Düsseldorf
Locations (1):
- Frauenklinik der Heinrich Heine Universität, Düsseldorf, Germany

REFERENCES:
- See also: SUCCESS-Trial homepage — http://www.success-studie.de